CLINICAL TRIAL: NCT03317366
Title: Expanded Access to Provide ARQ 092 for the Treatment of Overgrowth Diseases and/or Vascular Anomalies With Genetic Alterations of the PI3K/AKT Pathway
Brief Title: Expanded Access to Provide ARQ 092 for the Treatment of Overgrowth Diseases and/or Vascular Anomalies
Status: No longer available | Type: Expanded Access
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Other Study IDs: ARQ 092 Expanded Access
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Proteus Syndrome; PIK3CA-Related Overgrowth Spectrum (PROS); Growth Disorders
Keywords: ARQ 092; ArQule; AKT; PIK3CA; Overgrowth; Congenital malformations
MeSH Terms: conditions — Proteus Syndrome; Growth Disorders; Hereditary Sensory and Autonomic Neuropathies; Congenital Abnormalities | interventions — Miransertib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: ARQ 092 — Open-label expanded access for ARQ 092 capsules

SUMMARY:
ARQ 092 is being investigated for patients with overgrowth diseases and/or vascular anomalies with genetic alterations of the PI3K/AKT pathway and may be available for patients who are ineligible for an ongoing ARQ 092 clinical trial or have other considerations that prevent access to ARQ 092 through an existing clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Severe overgrowth diseases and/or vascular anomalies with confirmed somatic genetic alterations of PIK3CA or AKT
2. Are unable to participate in an ongoing ARQ 092 clinical trial
3. Willing and able to provide written, signed informed consent. In the case of a minor, a parent or legal guardian must sign an informed consent form.
4. Medically suitable for treatment with ARQ 092
5. Not eligible for any other available therapy for the diagnosed overgrowth disease and/or vascular anomaly with confirmed somatic genetic alterations of PIK3CA or AKT

Exclusion Criteria:

1. Currently enrolled in an ongoing clinical study of ARQ 092 or other investigational drug
2. Currently being treated with any inhibitor of the PI3K/AKT/mTOR pathway

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult